CLINICAL TRIAL: NCT06958783
Title: Detection of Changes in the Lipid Profile in Early-Stage Breast Cancer Patients Undergoing Neoadjuvant or Adjuvant Chemotherapy
Brief Title: Chemotherapy-induced Lipid Profile Changes in Women With Early Breast Cancer
Status: Completed | Type: Observational
Sponsor: Cancer center Stefan Kukura Hospital Michalovce (Other)
Collaborators: Pavol Jozef Safarik University (Other)
Responsible Party: Sponsor
Other Study IDs: ONKOMi-Breast cancer study-23
Record Dates: First submitted 2025-04-27; First posted 2025-05-06 (Actual); Last update posted 2025-05-30 (Actual); Status verified 2025-05

CONDITIONS: Breast Neoplasms; Lipid Profile; Dyslipidemia
Keywords: early-stage breast cancer; chemotherapy; cardiovascular risk factor
MeSH Terms: conditions — Breast Neoplasms; Dyslipidemias

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum samples collected for the analysis of lipid profiles, including measurements of total cholesterol (TC), triglycerides (TG), low-density lipoprotein cholesterol (LDL-C), and high-density lipoprotein cholesterol (HDL-C)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Female patients with early-stage breast cancer receiving neoadjuvant or adjuvant chemotherapy.: The cohort consists of adult female patients with newly diagnosed early-stage invasive breast cancer (stage IB-IIIB) scheduled to receive standardized neoadjuvant or adjuvant chemotherapy.
  Interventions: Other: Blood lipid monitoring in breast cancer patients during chemotherapy

INTERVENTIONS:
Other: Blood lipid monitoring in breast cancer patients during chemotherapy — This intervention is distinguished by its prospective design, enrollment of a clearly defined cohort of adult female patients with newly diagnosed early-stage breast cancer (stage IB-IIIB), administration of a uniform chemotherapy regimen (doxorubicin, cyclophosphamide, paclitaxel), and standardized monitoring of fasting lipid profiles at four precisely scheduled timepoints: pre-chemotherapy, pre-paclitaxel, post-paclitaxel, and three months post-chemotherapy completion

SUMMARY:
Detection of changes in the lipid profile in early-stage breast cancer patients undergoing neoadjuvant or adjuvant chemotherapy with doxorubicin, cyclophosphamide, and paclitaxel.

DETAILED DESCRIPTION:
Despite the development of highly effective antitumor therapies over the past two decades (e.g., targeted therapy, immunotherapy), chemotherapy regimens including anthracyclines, taxanes, and cyclophosphamide continue to represent a fundamental component of treatment algorithms for early breast cancer, particularly in human epidermal growth factor receptor 2 (HER2)-positive and triple-negative breast cancer (TNBC). While the cardiotoxicity of anthracyclines is well established and routinely monitored by echocardiography, changes in lipid profiles induced by cytotoxic chemotherapy have primarily been reported in retrospective studies with heterogeneous patient populations and measurement protocols.

This prospective, single-center study was designed to evaluate changes in lipid parameters in patients with early-stage breast cancer undergoing neoadjuvant or adjuvant chemotherapy with doxorubicin, cyclophosphamide, and paclitaxel.

ELIGIBILITY:
Inclusion Criteria:

Female patients with newly diagnosed breast cancer, stage IB-IIIB, assigned to receive neoadjuvant or adjuvant chemotherapy.

Histologically confirmed invasive adenocarcinoma of the breast, including hormone receptor-positive, HER2-positive (human epidermal growth factor receptor 2), or triple-negative breast cancer.

Chemotherapy regimen based on doxorubicin, cyclophosphamide, and paclitaxel.

Completion of all planned neoadjuvant or adjuvant chemotherapy cycles.

Availability of complete lipid profile data at all required timepoints.

Exclusion Criteria Prior breast cancer treatment (surgery, chemotherapy, radiotherapy, or systemic therapy).

Ongoing or prior treatment with hypolipidemic (lipid-lowering) medications.

Incomplete chemotherapy regimen (interrupted or prematurely terminated cycles).

Presence of distant metastatic disease at diagnosis.

Missing or incomplete lipid profile data.

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult female patients with newly diagnosed, histologically confirmed early-stage invasive breast cancer (stages IB-IVA) assigned to receive standardized neoadjuvant or adjuvant chemotherapy with doxorubicin, cyclophosphamide, and paclitaxel, treated at a single center.
Sampling Method: Non-Probability Sample
Enrollment: 56 (Actual)
Dates: Start 2023-03-05 (Actual); Primary Completion 2025-02-28 (Actual); Study Completion 2025-02-28 (Actual)

PRIMARY OUTCOMES:
Change in fasting lipid profile parameters (TC, TG, LDL-C, HDL-C) during and after chemotherapy | From enrollment (1-3 days prior to chemotherapy initiation) through three months after completion of chemotherapy.
  Evaluation of dynamic changes in fasting serum levels of total cholesterol (TC), triglycerides (TG), low-density lipoprotein cholesterol (LDL-C), and high-density lipoprotein cholesterol (HDL-C) at predefined timepoints during neoadjuvant or adjuvant chemotherapy and at three months after chemotherapy completion.

SECONDARY OUTCOMES:
Correlation of lipid profile changes with menopausal status and body mass index (BMI) | From enrollment (1-3 days prior to chemotherapy initiation) through three months after completion of chemotherapy.
  Assessment of the association between dynamic changes in fasting lipid parameters (TC, TG, LDL-C, HDL-C) and patients' menopausal status and body mass index (BMI) measured at baseline. The analysis aims to explore potential modifiers of chemotherapy-induced lipid alterations.

CONTACTS AND LOCATIONS:
Locations (1):
- Oncology Center, Štefan Kukura Hospital, Penta Hospitals, Michalovce, Michalovce, Slovakia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Rusinova L, Medvedieva J, Santova Z, Kozarova M. Prospective evaluation of chemotherapy-induced dyslipidemia in early breast cancer: implications for cardiovascular risk. Front Oncol. 2026 Jan 12;15:1677835. doi: 10.3389/fonc.2025.1677835. eCollection 2025. PMID 41602405